CLINICAL TRIAL: NCT04093635
Title: Role of Negative Pressure Wound Therapy in the Management of Diabetic Foot Ulcers
Brief Title: Negative Pressure Wound Therapy in the Management of Diabetic Foot Ulcers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ibrahim Sayed, Vascular Surgery Department, Assiut University, Assiut University
Other Study IDs: VAC in DFUs
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Those patients that will be treated by NPWT.
  Interventions: Device: Negative Pressure Wound Therapy
- Group II: Those patients will be treated with standard saline moist wound care and dressing.
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — VAC was applied by placing sterile pads in two layers with a 16Fr Ryle's tube placed between the two layers and then the wound was sealed by a sterile transparent polyurethane sheet. The tube was connected to a wall-mounted suction device and the pressure will be set at -125 mmHg Mode of NPWT. This dressing will be changed every 72 hrs

SUMMARY:
Role of Negative Pressure Wound Therapy in the Management of Diabetic Foot Ulcers

• The aim of this study will be to assess negative pressure wound therapy in treating diabetic foot ulcers.

DETAILED DESCRIPTION:
Diabetic Foot ulcers are a major cause of admission in diabetic patients, and comprise a disproportionately high number of hospital days because of multiple surgical procedures and prolonged length of stay in Hospital.

The improvement in diabetes therapy and the reinforcement of guidelines have reduced the amputation rate. The approach to diabetic foot ulcers has allowed the availability of several medical options to ensure the best local condition and wound healing.

Negative-pressure wound therapy is a non-invasive therapy system that employs a controlled negative pressure using a vacuum device to promote wound healing by removing fluid from open wounds through a sealed dressing or a foam dressing connected to a container.

An earlier study has shown that NPWT reduced the need for subsequent amputations in a 6-month follow-up period. This reflects the importance of this device in management of DFUs and prevents its complications.

As most of the diabetic wounds present with infection, the success of NPWT is still highly dependent upon the adequacy of surgical debridement and antimicrobial coverage.

NPWT provides a moist wound environment ideal for re-epithelialization, growth factor action, angiogenesis, and granulation promotion.

Edema reduction produced by NPWT decreases interstitial pressure and positively promoting wound vessel formation and improving wound circulation and lymphatic drainage, increasing the availability of nutrients, oxygen and antibiotic therapy in the wound area. Some studies showed that NPWT promotes an improvement of balance between proteases and their inhibitors and influences cytokine modulation and promotes a positive wound environment.

Accurate classification of diabetic foot ulcers according to Wagner's classification of ulcers is essential for inter-clinician communication, assessment of healing tendency during management by NPWT.

ELIGIBILITY:
Inclusion Criteria:

* Acute and chronic diabetic wounds, pressure ulcers.
* Wagener's Grade I superficial diabetic ulcer.
* Wagener's Grade II after surgical debridement and an appropriate antibiotic therapy.
* Ischemic wounds after revascularization.

Exclusion Criteria:

* - Wagener's Grade III, osteomyelitis and Charcot's joint septic arthritis.
* Wagener's Grade IV, localized gangrene e.g. toe ,heel.
* Wagener's Grade V, extensive gangrene involving the whole foot.
* Septicemia. .
* Gas forming organism.
* Wounds resulting from venous insufficiency.
* Peripheral vascular disease (absent distal pulse).
* Patients being treated with corticosteroids, immunosuppressive drugs or chemotherapy
* Any other serious pre-existing cardiovascular, pulmonary and immunological disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients diagnosed as DFU from November 2019 to November 2020 at Assiut University Hospital.
  The patients will divide into two groups:
  Group I: Those patients that will be treated by NPWT. Group II: Those patients will be treated with standard saline moist wound care and dressing.
  Each group consists of 20 patients.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Management of diabetic foot ulcers. | one year
  Assessment role of negative pressure wound therapy in treating diabetic foot ulcers.

REFERENCES:
- [Background] Iheozor-Ejiofor Z, Newton K, Dumville JC, Costa ML, Norman G, Bruce J. Negative pressure wound therapy for open traumatic wounds. Cochrane Database Syst Rev. 2018 Jul 3;7(7):CD012522. doi: 10.1002/14651858.CD012522.pub2. PMID 29969521
- [Background] Liu S, He CZ, Cai YT, Xing QP, Guo YZ, Chen ZL, Su JL, Yang LP. Evaluation of negative-pressure wound therapy for patients with diabetic foot ulcers: systematic review and meta-analysis. Ther Clin Risk Manag. 2017 Apr 18;13:533-544. doi: 10.2147/TCRM.S131193. eCollection 2017. PMID 28458556
- [Background] James SMD, Sureshkumar S, Elamurugan TP, Debasis N, Vijayakumar C, Palanivel C. Comparison of Vacuum-Assisted Closure Therapy and Conventional Dressing on Wound Healing in Patients with Diabetic Foot Ulcer: A Randomized Controlled Trial. Niger J Surg. 2019 Jan-Jun;25(1):14-20. doi: 10.4103/njs.NJS_14_18. PMID 31007506
- [Background] Borys S, Hohendorff J, Koblik T, Witek P, Ludwig-Slomczynska AH, Frankfurter C, Kiec-Wilk B, Malecki MT. Negative-pressure wound therapy for management of chronic neuropathic noninfected diabetic foot ulcerations - short-term efficacy and long-term outcomes. Endocrine. 2018 Dec;62(3):611-616. doi: 10.1007/s12020-018-1707-0. Epub 2018 Aug 11. PMID 30099674
- [Background] Hu X, Lian W, Zhang X, Yang X, Jiang J, Li M. Efficacy of negative pressure wound therapy using vacuum-assisted closure combined with photon therapy for management of diabetic foot ulcers. Ther Clin Risk Manag. 2018 Oct 25;14:2113-2118. doi: 10.2147/TCRM.S164161. eCollection 2018. PMID 30498354